# Informed Consent Form

Title: Improving Clinical Trial Recruitment and Outcome Measures in Bullous Pemphigoid

NCT # NCT04728854

Date: 06/12/2023

## You Are Being Asked to Be in a Research Study Concise presentation of key concepts

You are being asked to be in a research study. A research study is designed to answer a scientific question. If you agree to be in the study you will be one of 45 people who are being studied, at Emory.

## Why is this study being done?

This study is being done to answer the question: How to improve clinical trial outcome measures for patients with bullous pemphigoid. You are being asked to be in this research study to help define appropriate measurements over time while on treatment and to assess the use of teledermatology for follow-up visits.

## Do you have to be in the study?

It is your decision to be part of this research study. You do not have to be in it. Your choice will not affect your access to medical care for your condition. Before you make your decision, you should take time to learn about the study.

## What do I have to do if I choose to participate in this study?

If you are eligible and want to be part of the study, you will participate for 6 months which will include 5 study visits, four of which will be at your place of residence. The researchers will ask you to do the following: Basic clinical evaluation with pemphigoid scoring, quality of life surveys and photographs. Some of these procedures will be paid for by the study.

## How is this study going to help you?

If you are in the study, you will be helping the researchers answer the study question, How to improve clinical trial design for patients who suffer with bullous pemphigoid.

## What are the risks or discomforts I should know about before making a decision?

The study will take time. All studies have some risks. Some risks are relatively small, like being bored or losing time. Some are more serious – for this study, these include loss of privacy, and breach of confidentiality. A full list of expected risks, their frequency and severity are in the "What are the possible risks and discomforts?" section of this document.

#### Alternatives to Joining This Study

Since this is not a treatment study, the alternative is not to participate

#### Costs

You WILL not have to pay for any of the study procedures, in particular those that are not covered by your medical insurance.

#### What Should I Do Next?

Read this form, or have it read to you. Make sure the study doctor or study staff explains the study to you. Ask questions (e.g., about exact time commitment, about unfamiliar words, more details on specific procedures, etc.) Make sure you understand Take time to consider this, and talk about it with your which parts of the are research and which are standard care that you would have even if you did not join the study. family and friends.

Version Date: 09/07/2021

 IRB Form 06162020



# Emory University Consent to be a Research Subject / HIPAA Authorization

<u>Title</u>: Improving Clinical Trial Recruitment and Outcome Measures in Bullous Pemphigoid

IRB #: STUDY00001274

Principal Investigator: Ron Feldman, MD, PhD

**Sponsor:** NIH/NIAMS

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form, you will not give up any legal rights.

A description of this clinical trial is available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

## What is the purpose of this study?

The purpose of this study is to define appropriate outcome measures for proper clinical trial design in patients with bullous pemphigoid

#### What will I be asked to do?

You will be asked to view a video that will tell you about the study.

You will be asked to participate in a screening/baseline visit which will include taking photographs, month 1, 2, 3, 4 and a follow up visit at month 8 - 10. Visits will be conducted remotely via telehealth where you will be asked to take and provide self-captured photographs.

If you were referred to the Emory Autoimmune Blistering Disease Clinic while you were hospitalized, you authorize the use of consultation photographs to be utilized as study data.

Surveys to be Completed by all Patients enrolled in study:

Demographic: A questionnaire that asks your age, gender, race, and education

 IRB Form 06162020



- BPDAI: Bullous pemphigoid disease area index; An evaluation of your skin and mucosal membranes for blisters, redness, and pigment changes of your skin involved with bullous pemphigoid
- ItchyQol: A questionnaire about itch and how it affects your quality of life
- ItchyQuant:A questionnaire about itch and how it affects your quality of life
- ABQOL: A questionnaire about how your blisters affect your quality of life
- TABQOL: A questionnaire about how treatment for your bullous pemphigoid affects your quality of life

## Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may be still be used for this study.

## What are the possible risks and discomforts?

This is a minimal risk study but it is possible you could experience some psychological discomfort with the questions on the surveys. You did not have to answer any question that you do not want to answer. There is also a risk of breach of confidentiality.

## Will I benefit directly from the study?

This study is not designed to benefit you directly. Your bullous pemphigoid may improve while you are in this study but it may not, and it may even get worse. This study is designed to learn more about appropriate measurements over time and potential use of remote monitoring of patients in clinical research for bullous pemphigoid. The study results may be used to help others in the future.

## Will I be compensated for my time and effort?

You will get \$50.00 gift card at the screening/baseline visit and a \$30.00 gift card at each completed subsequent visit. If you do not finish the study, we will compensate you for the visits you have completed. You will get \$200.00 total, if you complete all study visits.

## What are my other options?

If you decide not to enter this study, there is care available to you outside of this research study. The study doctor will discuss these with you. You do not have to be in this study to be treated for bullous pemphigoid.

## How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

Study records can be opened by court order. They also may be provided in response to a subpoena or a request for the production of documents.

Certain offices and people other than the researchers may look at study records which include photographs. Government agencies and Emory employees overseeing proper study conduct may look at your study records. These offices include the Office for Human Research Protections, the funder(s), the Emory Institutional Review Board, the Emory Office of Research Compliance. Study funders may also look at your study records. Emory

Version Date: 09/07/2021




will keep any research records we create private to the extent we are required to do so by law. A study number rather than your name will be used on study records wherever possible. Your name and other facts that might point to you will not appear when we present this study or publish its results.

## **Storing and Sharing your Information**

De-identified data from this study (data that has been stripped of all information that can identify you), may be placed into public databases where, in addition to having no direct identifiers, researchers will need to sign data use agreements before accessing the data. We will remove or code any personal information that could identify you before your information is shared. This will ensure that, by current scientific standards and known methods, it is extremely unlikely that anyone would be able to identify you from the information we share. Despite these measures, we cannot guarantee anonymity of your personal data.

Your data [and specimens] from this study may be useful for other research being done by investigators at Emory or elsewhere. To help further science, we may provide your deidentified data and/or specimens to other researchers. If we do, we will not include any information that could identify you. If your data or specimens are labeled with your study ID, we will not allow the other investigators to link that ID to your identifiable information.

We will use your sample and data only for research. We will not sell them. However, the results of this research might someday lead to the development of products (such as a commercial cell line, a medical or genetic test, a drug, or other commercial product) that could be sold by a company. You will not receive money from the sale of any such product.

In general, we will not give you any individual results from the study of the samples you give us. If we find something of urgent medical importance to you, we will inform you, although we expect that this will be a very rare occurrence.

#### In Case of Injury

If you believe you have become ill or injured from this research, you should contact Dr. Feldman at telephone number . You should also let any health care provider who treats you know that you are in a research study.

If you get ill or injured from being in the study, Emory will help you to get medical treatment. Neither Emory nor the sponsor have set aside money to pay for this medical treatment. Your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurance does not pay, then you will have to pay these costs.

For Emory, the only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory employee. "Negligence" is the failure to follow a standard duty of care. You do not give up any legal rights you may have by being in this study, including any right to bring a claim for negligence.

 IRB Form 06162020 Version Date: 09/07/2021



## **Costs**

There will be no costs to you for participating in this study, other than basic expenses like transportation. You will not be charged for any of the research activities. If the study procedures result in any medical complications that would not fall under "injury" as discussed above, the cost of treatment for those complications may be charged to you or your insurance.

The actual amount that you have to pay depends on whether or not you have health insurance and whether or not that insurance will pay for any research study costs. Generally, insurance companies will not pay for items and services that are required just for a research study. Some insurance companies will not pay for regular medical treatment or treatment for complications if you are in a study. How much you will have to pay for any co-payments, deductibles or co-insurance depends on your plan. Emory and the sponsor will not pay for these costs.

It is a good idea to contact your insurance provider and tell them you want to be in this research study. Ask them what they will pay for and what they will not pay for. You can also ask the study team for help in figuring out what you will have to pay.

If you do not have insurance, Emory will review your case as part of its program for low-income patient care. The standard policies of that program will apply. The program will figure out if you have to pay any costs for taking part in the study and what those costs will be.

## Withdrawal from the Study

You have the right to leave a study at any time without penalty.

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

#### **Authorization to Use and Disclose Protected Health Information**

The privacy of your health information is important to us. As part of this study, we will be requesting health care entities who are covered by the Health Insurance Portability and Accountability Act and regulations (HIPAA) to provide us with health information that identifies you ("individually identifiable health information" or "IIHI"). Because the health care entities are covered by HIPAA, we must have your authorization to obtain your IIHI from them. However, the researchers who get your IIHI from the health care entities are not covered by HIPAA. Once they receive your IIHI from the health care entities, they will put it in a separate research record that is not a part of your medical record. IIHI placed in the separate research record is not be covered by HIPAA.

## **Purpose of this Authorization:**

By signing this form, you give us permission to get your IIHI from health care entities and to use and share your IIHI as described in this document. You do not have to sign this form. If you do not sign this form, then you may not participate in the research study.

Version Date: 09/07/2021

 IRB Form 06162020



#### No Provision of Treatment

There is no research-related treatment involved in this study. You may receive any non-research related treatment whether or not you sign this form.

## IIHI that Will be Used/Disclosed:

The IIHI that we will use or share for the research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.
- Photographs taken by research personnel.
- Self-Captured Photographs.

## Purposes for Which Your IIHI Will be Used/Disclosed:

We will use and share your IIHI for the conduct and oversight of the research study. Once we have your IIHI we will keep it in a separate research record that will be used for the conduct of the study. If you leave the study, we may use your IIHI to determine your vital status or contact information.

## Use and Disclosure of Your IIHI That is Required by Law:

We will use and disclose your IIHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your IIHI. These include subpoenas or court orders.

#### People Who will Use/Disclose Your IIHI:

The following people and groups will use and disclose your IIHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your IIHI to conduct the study.
- The Principal Investigator and research staff will share your IIHI with other people and groups to help conduct the study or to provide oversight for the study. This includes sharing your IIHI with people and groups at other sites who are helping conduct the study.
- The following people and groups will use your IIHI to make sure the research is done correctly and safely:
  - Emory offices that are part of the Human Research Participant Protection Program and those that are involved in study administration. These include the Emory IRB, the Emory University and Healthcare Compliance Offices, and the Emory Office for Clinical Research.
  - Public health agencies.
  - Research monitors and reviewer.
  - Accreditation agencies.
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens, your IIHI may be shared with that new institution and their oversight offices.

 Version Date: 09/07/2021



## **Expiration of Your Authorization**

Your IIHI will be used until this research study ends.

#### **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your IIHI. If you want to do this, you must contact the study team at:

At that point, the researchers would not collect any more of your IIHI. But they may use or disclose the information you already gave them as described in this Authorization. If you revoke your authorization you will not be able to stay in the study.

## Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. HIPAA does not apply to research that does not include treatment that is billed to insurers or government benefit programs. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them.

To maintain the integrity of this research study, you generally will not have access to your IIHI related to this research until the study is complete. When the study ends, and at your request, you generally will only have access to your IIHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. You will not have a right of access to IIHI kept in a separate research record used only for research purposed. If it is necessary for your health care, your health information will be provided to your doctor.

We may remove identifying information from your IIHI. Information without identifiers is not subject to HIPAA and may be used or disclosed with other people or organizations for purposes besides this study.

#### **Contact Information**

Contact Dr. Ron Feldman at

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or
- if you have questions, or concerns about the research

Contact the Emory Institutional Review Board at

- if you have questions about your rights as a research participant.
- if you have complaints about the research or an issue you rather discuss with someone outside the research team.

You may also let the IRB know about your experience as a research participant through our Research Participant Survey at https://tinyurl.com/ycewgkke.

Version Date: 09/07/2021



# **Consent and Authorization**

| TO BE FILLED OUT BY SUBJECT Please print your name, sign, and date below if you agree to be in the and authorization form, you will not give up any of your legal rights. We keep. | nis research stud | |
|---|---|---|
| Name of Subject | | |
| Signature of Subject (18 or older and able to consent) | Date | Time |
| TO BE FILLED OUT BY STUDY TEA | M ONLY | |
| Name of Person Conducting Informed Consent Discussion | | |
| Signature of Person Conducting Informed Consent Discussion | <br>Date | Time |